CLINICAL TRIAL: NCT02224482
Title: Randomized Clinical Trial of an Online Multimedia Program to Boost Coping & Function for Prostate Cancer Survivors
Brief Title: Trial of an Online Multimedia Program to Boost Coping & Function for Prostate Cancer Survivors (PROGRESS)
Acronym: PROGRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1R01CA158019 (NIH); R01CA158019 (NIH)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Helio Progress

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Print materials
- Intervention Group (Active Comparator): PROGRESS
  Interventions: Behavioral: PROGRESS

INTERVENTIONS:
Behavioral: PROGRESS — PROGRESS is a multimedia website designed to help prostate cancer survivors.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to test how well an online program designed to help prostate cancer survivors cope with changes caused by their cancer or treatment works compared to standard print educational materials from the National Cancer Institute (NCI).

DETAILED DESCRIPTION:
This study involves the development and evaluation of a comprehensive and innovative multimedia program designed to facilitate the post-treatment transition into survivorship. The design of the intervention, the PRostate Cancer Online Guide and Resources for Electronic Survivorship Service (PROGRESS), is theoretically based on the team's Cognitive-Social Health Information Processing Model.

PROGRESS focuses on promoting adaptive coping within four key post-treatment domains: 1) Physical Dysfunction (e.g., physical symptoms); 2) Emotional Well- Being (e.g., fear of recurrence); 3) Interpersonal Concerns (e.g., sexual intimacy issues); and 4) Practical Barriers (e.g., medical follow-up challenges). Content for these domains are organized in a virtual resource center and will consist of: 1) provision of related information through text, graphics, voice overs, and animation; 2) videos of health care experts answering frequently asked questions; 3) videos of prostate cancer survivors describing their experiences and modeling competencies and coping strategies; and 4) skills training to improve communication between prostate cancer survivors and family and healthcare providers. Program content has been developed through literature and evidence-based content review, expert input, and input from multi-ethnic survivor focus groups. To ensure adequate and appropriate program content and optimal functionality, an iterative process of review, revision, and user and usability testing has been employed.

Intervention efficacy will be evaluated through a two-arm, prospective randomized controlled trial. A total of 600 patients (200 from Fox Chase Cancer Center, 200 from the Cancer Institute of New Jersey, and 200 from Icahn School of Medicine at Mount Sinai) will complete the study. Data will be collected at baseline, and at 1-, 3- and 6- months follow-up.

The primary outcome variable will be use of adaptive coping, and secondary outcome variables will include use of maladaptive coping, disease-specific quality of life, vitality/energy, physical quality of life, cancer-related intrusive thoughts, emotional quality of life, fear of recurrence, bother from physical dysfunctions, satisfaction with communication in medical interactions, satisfaction with cancer-related with family/friends, marital problems, and practical concerns . A theory-based test of mediators of intervention effects (i.e., self-efficacy for the survivorship phase, confidence in ability to manage symptoms related to prostate cancer, perceived information utility), and moderators (i.e., demographics, comorbid conditions, monitoring style, affect) will also be performed.

The proposed research will be the first Randomized Controlled Trial to evaluate a comprehensive and highly disseminable and self-sustaining intervention for facilitating post-treatment adaptation among early-stage Pca survivors. In addition, use of and usability, accessibility, and satisfaction with PROGRESS will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Received a diagnosis of localized disease confined to the prostate, with no regional lymph node or distant metastasis (stages T1, T1a, T1b, T2, T2a, T2b; T2c [3]);
* Within one year completion of either radical prostatectomy or radiation therapy(external beam radiation therapy or brachytherapy);
* Have access to a personal computer with Internet access (either in home or at a community center);
* 18 years of age or older;
* Able to communicate in English
* Able to give consent

Exclusion Criteria:

* Unable to use a computer
* Unable to communicate in English

Exclusion Criteria:

* unable to use a computer
* unable to communicate in English

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Miller, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (3):
  - Rutgers Cancer Insititute of New Jersey, Somerset, New Jersey
  - Icahn School of Medicine at Mt Sinai, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Marziliano A, Diefenbach MA, Hudson SV, Tagai EK, Handorf EA, Bator A, Miller SM. Demographic and Psychosocial Characteristics Associated With Use of a Prostate Cancer Survivorship Website: Implications From a Multisite Randomized Controlled Trial. J Med Internet Res. 2022 Mar 21;24(3):e27890. doi: 10.2196/27890. PMID 35311678

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention Group
Started | 214 | 217
Completed | 63 | 57
Not Completed | 151 | 160

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention Group | Total
Number analyzed (Participants) | 214 | 217 | 431
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (7.5) | 63.8 (6.7) | 63.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 214 | 217 | 431
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Different counts due to missing data
  Participants
    Non-Hispanic White | 143 | 160 | 303
    Black | 51 | 40 | 91
    Other | 18 | 17 | 35
    Unknown | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 214 | 217 | 431
PSA at diagnosis (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 8.6 (10.7) | 14.0 (49.0) | 11.4 (35.6)
Prostate cancer treatment completed [Count of Participants; unit: Participants] — Population: Counts different due to missing data
  Participants
    Surgery Only: number analyzed (Participants) | 212 | 213 | 425
    Surgery Only | 131 | 130 | 261
    Radiation Only: number analyzed (Participants) | 212 | 213 | 425
    Radiation Only | 50 | 59 | 109
    Other (multiple treatments): number analyzed (Participants) | 212 | 213 | 425
    Other (multiple treatments) | 31 | 24 | 55

OUTCOME MEASURES:

1. Primary Outcome: Adaptive Coping
Description: Adaptive coping was measured with the Cancer Coping Questionnaire. The total score from the Cancer Coping Questionnaire is a mean scale. There were a total of 14 items, each with a Likert-type 4-point scale, with 1 being the minimum value and 4 being the maximum value. A higher score indicated greater coping ability (i.e., better outcome).
Time Frame: Change in coping from baseline to six months
Population: Data provided for participants with six month data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 106 | 103
score on a scale | -0.089 (0.559) | -0.013 (0.602)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .9634, Mixed Models Analysis

2. Secondary Outcome: Physical Functioning - Urinary Incontinence
Description: This will be measured using the Urinary Incontinence Scale from the Expanded Prostate Cancer Index Composite - Short Form (EPIC 26-SF), a 26 item shortened version of EPIC, a 61 item questionnaire for assessing urinary, bowel, sexual, and hormonal dysfunction and distress/bother in prostate cancer patients. The scale had four items, each with a Likert-type 4- or 5-item scale, with 1 being the minimum and 4 or 5 being the maximum. These scores were then recoded to a 0 to 100 scale, with higher scores indicating less urinary incontinence (i.e., better outcome).
Time Frame: Change from baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 101 | 96
score on a scale | 9.240 (19.671) | 10.750 (21.933)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .5214, Mixed Models Analysis

3. Secondary Outcome: Physical Functioning - Urinary Irritation
Description: This will be measured using the Urinary Irritation Scale from the Expanded Prostate Cancer Index Composite - Short Form (EPIC 26-SF), a 26 item shortened version of EPIC, a 61 item questionnaire for assessing urinary, bowel, sexual, and hormonal dysfunction and distress/bother in prostate cancer patients. The scale had four items, each with a Likert-type 4- or 5-item scale, with 1 being the minimum and 4 or 5 being the maximum. These scores were then recoded to a 0 to 100 scale, with higher scores indicating less urinary irritation (i.e., better outcome).
Time Frame: Change from baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 100 | 94
score on a scale | 10.063 (17.200) | 7.979 (16.660)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .4875, Mixed Models Analysis

4. Secondary Outcome: Physical Functioning - Bowel
Description: This will be measured using the Bowel Scale from the Expanded Prostate Cancer Index Composite - Short Form (EPIC 26-SF), a 26 item shortened version of EPIC, a 61 item questionnaire for assessing urinary, bowel, sexual, and hormonal dysfunction and distress/bother in prostate cancer patients. The scale had six items, each with a Likert-type 4- or 5-item scale, with 1 being the minimum and 4 or 5 being the maximum. These scores were then recoded to a 0 to 100 scale, with higher scores indicating less bowel problems (i.e., better outcome).
Time Frame: Change from baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 102 | 97
score on a scale | 1.479 (13.330) | 3.119 (14.847)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .7938, Mixed Models Analysis

5. Secondary Outcome: Physical Functioning - Sexual Functioning
Description: This will be measured using the Sexual Functioning Scale from the Expanded Prostate Cancer Index Composite - Short Form (EPIC 26-SF), a 26 item shortened version of EPIC, a 61 item questionnaire for assessing urinary, bowel, sexual, and hormonal dysfunction and distress/bother in prostate cancer patients. The scale had six items, each with a Likert-type 4- or 5-item scale, with 1 being the minimum and 4 or 5 being the maximum. These scores were then recoded to a 0 to 100 scale, with higher scores indicating less sexual problems (i.e., better outcome).
Time Frame: Change from baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 98 | 96
score on a scale | 4.793 (19.829) | 3.046 (21.402)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .6765, Mixed Models Analysis

6. Secondary Outcome: Interpersonal Concerns - Medical Interactions
Description: Satisfaction with communication in medical interactions will be assessed with the medical interactions scale from the Cancer Rehabilitation Evaluation System (CARES): difficulty communicating with the medical team, and problems obtaining information from the medical team. The minimum value is 0 and the maximum value is 4. A higher score means patients had worse medical interactions (i.e., worse outcome).
Time Frame: Change from baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 103 | 96
score on a scale | -0.311 (2.783) | -0.531 (2.554)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .7061, Mixed Models Analysis

7. Secondary Outcome: Interpersonal Concerns - Marital Interactions
Description: Satisfaction with marital communication will be assessed from the marital problems scale from the Cancer Rehabilitation Evaluation System (CARES). The minimum value is 0 and the maximum value is 4. A higher score means more marital problems (i.e., worse outcome).
Time Frame: Change from baseline to six months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Intervention Group
Number analyzed (Participants) | 95 | 88
score on a scale | -0.042 (3.956) | 0.182 (3.358)
Statistical Analysis 1: Comparison: Control vs Intervention Group; Test type: Superiority; p = .7593, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each participant over a 6 month period through 6-month follow-up.
Description: No adverse events anticipated in low-risk behavioral trial.
Arm/Group | Control | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/214 | 0/217
Serious Adverse Events (participants affected / at risk) | 0/214 | 0/217
Other Adverse Events (participants affected / at risk) | 0/214 | 0/217

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT02224482/Prot_SAP_000.pdf